CLINICAL TRIAL: NCT06199557
Title: A Phase 1/2 Multicenter Open-label Study to Investigate Treatment of Hydroxyurea in Combination With Valproic Acid (VPA), or 6- Mercaptopurine in Combination With VPA in Patients With AML or HR-MDS Unfit for Standard Therapy
Brief Title: A Study to Investigate Treatment of HU and VPA, or 6-MP and VPA in Unfit AML/HR-MDS Patients
Acronym: HUVAMER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUVPA_6MPVPA
Record Dates: First submitted 2023-12-12; First posted 2024-01-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia, Adult; Myelodysplastic Syndromes, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Hydroxyurea; Valproic Acid; Epilim; Mercaptopurine

STUDY DESIGN:
Intervention Model Description: This a two-part, open-label phase 1/2 study that will include clinical sites in Norway and other Nordic countries. The study consists of part A and part B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxyurea (HU) + Valproic Acid (VPA) part 1 (Active Comparator): Combination treatment 1 (T1): hydroxyurea + valproic acid, combination treatment 2 (T2): 6-mercaptopurine + valproic acid.
  Each patient enrolled will receive at least one cycle with T1: hydroxyurea and valproic acid. The 1st cycle in the study always constitutes of hydroxyurea (1000 mg twice a day) plus valproic acid (300 mg + 600 mg) for 14 days; then 14 days with no medication.
  Each cycle duration is 28 days. Patients who do not experience clinical benefit after 1st cycle, or experience unacceptable and unmanageable toxicity after 1st cycle, will not be eligible to continue on this regimen and they will be allocated to treatment combination 2. T2 constitutes of 6-mercaptopurine ( 50 mg once a day) plus valproic acid 300 mg + 600 mg ) for 14 days; followed by 14 days with no medication. Each cycle duration is 28 days.
  Interventions: Drug: Hydroxyurea, Hydroxycarbamide; Drug: Valproic acid; Drug: 6-Mercaptopurine (6-MP)
- Hydroxyurea (HU) + Valproic Acid (VPA) part 2 (Active Comparator): Part B consists of two cohort expansions where the setup is identical to part A: one for HU + VPA and one for 6-MP + VPA, 16 patients in each, in total 32 new patients.
  In part B the same principles will apply for response, withdrawal and allocation from HU+ VPA to 6-MP + VPA. The treatment duration in all arms can last to up 6 cycles in total. Each cycle duration is 28 days.
  Interventions: Drug: Hydroxyurea, Hydroxycarbamide; Drug: Valproic acid; Drug: 6-Mercaptopurine (6-MP)

INTERVENTIONS:
Drug: Hydroxyurea, Hydroxycarbamide — Hydroxyurea (HU/hydroxycarbamide) is a hydroxylated analogue of urea which prevents DNA synthesis by inhibiting the activity of ribonucleotide reductase (RNR). HU has been used to treat a variety of diseases. As an antineoplastic drug, HU has some advantages. It may be used by ambulatory patients and has relatively few side effects, which are relieved almost immediately after withdrawal of the drug. The drug is readily absorbed from the gastrointestinal tract following oral administration. At present, HU has an important role as standard of care for treating hyperleukocytosis in chronic and acute myeloid leukemia.
  Other Names: Hydroxyurea Medac
Drug: Valproic acid — Valproic acid (VPA) has been used clinically as an anticonvulsant and mood-stabilizing drug. During the last two decades, VPA has been described as a histone deacetylase (HDAC) inhibitor and gained increased interest for use in cancer therapy. VPA is administered orally with available routine measurements of serum levels and has a low toxicity profile.
  Other Names: Orfiril Long depot; Belvo; Depakote; Dyzantil; Convulex; Syonell; Epilim
Drug: 6-Mercaptopurine (6-MP) — In 1953, 6-MP was an approved antileukemic agent resulting in remissions in children with acute lymphocytic leukemia (ALL). After adding 6-MP to methotrexate and prednisolone in the treatment regimen, the one-year mean survival of children with ALL was increased from 29% to 50%. 6-MP, even about 70 years after its discovery, remains the standard maintenance therapy once the children are in complete remission.
  Other Names: Puri-Nethol

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and preliminary efficacy of the combination treatment of hydroxyurea capsules and valproic acid capsules, or the combination treatment of 6-mercaptopurine tablets and valproic acid capsules in male and female patients aged 18 years or older with acute myeloid leukemia or high- risk myelodysplastic syndrome.

The population to be studied is newly diagnosed AML patients who are considered unfit for standard induction chemotherapy, HR-MDS unfit/ineligible for standard treatment, and relapsed/refractory AML/HR-MDS patients who are considered unfit for standard therapy ,or are, for some reason, ineligible for another type of therapy. Clinically, hydroxyurea, valproic acid and 6-mercaptopurine are historically very well-known therapeutic agents with low toxicity profiles. The rationale for this study is that the combination of these drugs with low toxicity will be well tolerated in elderly AML patients with comorbidities, or lower performance status. This combination could have a beneficial therapeutic effect on overall survival and contribute to a better quality of life.

DETAILED DESCRIPTION:
This a two-part, open-label phase 1/2 study that will include clinical sites in Norway and other Nordic countries.

The study consists of part A and part B. Part A will run in Norway only. Part B will run in Norway and the Nordic countries.

Both part A and part B have two different treatment combinations (T), combination 1 and combination 2. Part B is a cohort expansion of part A (if part A proves to be positive).

Treatment combination 1 (T1): hydroxyurea + valproic acid. Treatment combination 2 (T2): 6-mercaptopurine + valproic acid.

Each patient enrolled in the trial will start and will receive at least one cycle with T1:

hydroxyurea and valproic acid. The first cycle in the study always constitutes of hydroxyurea (1000 mg twice a day) plus valproic acid (300 mg + 600 mg) for 14 days; this will be followed by a 14-day period with no medication. Each cycle duration is 28 days.

Patients who do not experience clinical benefit after the first cycle will not be eligible to continue on this regimen and they will be allocated to treatment combination 2. On the other hand, patients who do experience clinical benefit after cycle 1 with combination 1 (HU + VPA) will be further eligible to continue on this regimen/combination. However, patients on T1 will be withdrawn after consequent cycles, as soon as they do not meet the criteria for clinical benefit as defined by this protocol. Each patient who does not meet the criteria of clinical benefit after the first cycle with treatment combination 1 will switch to treatment combination 2 (T2). T2 constitutes of 6-mercaptopurine (50 mg once a day) plus valproic acid (300 mg + 600 mg) for 14 days; this will be followed by a 14-day period with no medication. Each cycle duration is 28 days. Patients will be further eligible to continue this regimen/combination for as long as they experience clinical benefit, otherwise they will be withdrawn from the study as soon as they do not meet the criteria for clinical benefit as defined by this protocol.

There will be 8 patients allocated for the treatment combination 1 with HU + VPA and up to 8 patients allocated for the treatment combination 2 with 6MP + VPA. For each of the two treatment combinations, if one or more patients, of 8, experience clinical benefit* the group will be expanded with 16 more patients in Part B. Part B consists of two cohort expansions where the setup is identical to part A, one for HU + VPA and one for 6MP + VPA, 16 patients in each, in total up to 32 new patients.

In part B, the same principles will apply for response, withdrawal and allocation from HU+ VPA to 6MP + VPA. Patients treated with combination 1, who do not experience clinical benefit or experience unacceptable, unmanageable toxicity after cycle 1, will not be eligible to continue on this regimen, and they will be allocated to combination 2. It is expected that cohort expansion of combination 2 will proceed slower than cohort expansion for combination 1.

If 5 or more patients of the total of 24 (part A (n=8) + part B (n=16)) experience clinical benefit, there will be considered a phase II/III expansion cohort for further effect assessment.

The treatment duration in all groups can last to up 6 cycles in total, each cycle lasts for 28 days. The rationale for the flow in the study aims to ensure that the patients do not undergo prolonged periods with excessive and ineffective treatment. Assessment of treatment response consecutively after each cycle will guide the treating physician to swiftly change the treatment combination or withdraw the patient from the study accordingly.

The switch to a second treatment combination as a part of the study ensures that more therapy options are available for, potentially, all patients who enroll in the trial.

The enrollment is stopped when 8+16 patients with HU +VPA are treated, or if 8+16 patients are treated with 6MP + VPA. Patients will switch over to 6MP +VPA, if lack of clinical benefit. Some dose modifications are allowed when indicated according to the protocol. At screening and during the study treatment, tumor debulking with HU + 6MP is required for 5 to 7 days to reduce WBC to less than 25×10*9/L (<20% blasts in the peripheral blood), before each cycle, HU + VPA, or 6MP + VPA. Tumor debulking with HU + 6MP may be repeated ahead of every cycle (for both treatment combinations), and in the treating physician's discretion, if the patient tolerates this.

The objectives of this study include:

* To determine the safety and tolerability of the treatment combinations of hydroxyurea + valproic acid, and 6-mercaptopurine + valproic acid administered at established clinical doses
* To establish the preliminary efficacy of the treatment combination of hydroxyurea and valproic acid administered at established clinical doses
* To establish the preliminary efficacy of the treatment combination of 6-mercaptopurine and valproic acid administered at established clinical doses
* To evaluate changes in patients performance status for baseline and during the study period

The adaptive study design is based on a Simon two-stage model of expanding cohorts. This model, tested in the TAPUR, DRUP and Impress-Norway studies, has been designed to effectively test a set of drugs using a minimum of number of patients (see also Chapter 9 on Statistics).

Each arm (A1, A2, B1 and B2) will be monitored using a Simon-like two-stage 'admissible' monitoring plan to identify patients with evidence of clinical benefit. Both arms in part A will enroll 8 participants, and will be considered positive if ≥1 patient show clinical benefit after at least 28 days on treatment (for each arm). In case of a positive part A (arm A1 and A2, separately), part B (arm B1 and B2, separately) will be initiated enrolling 16 additional participants in each arm into the cohort.

If there are 0 patients with "clinical benefit" (as defined by this protocol) among the first 8 participants in an arm, then the respective arm will not proceed to expansion. Otherwise, an additional 16 participants will be included in each cohort expansion (B1 and B2, respectively). Four or fewer responses out of 24 will suggest a lack of activity, while 5 or more responses will suggest that further investigation of the drug in a phase 3 clinical trial is warranted.

* Study duration: 5 years
* Treatment duration: up to 6 months for each treatment combination
* Visit frequency: every 7 days (if applicable, during the first cycle), thereafter every 28 days

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for the study only if all of the following criteria apply:

o Female or male, age 18 years or older

* Written informed consent
* Patients with Newly diagnosed AML, as defined by ELN 2022 criteria, or relapsed/refractory AML who: - are unfit, defined as HCT-CI ≥ 3, or - in the opinion of the investigator are not candidates for standard therapy or unlikely to tolerate or derive significant clinical benefit from standard therapy, or

  * the patient has declined standard therapy

Newly diagnosed HR-MDS, or relapsed/refractory HR-MDS who:

* are unfit, defined as HCT-CI ≥ 3, or
* in the opinion of the investigator are not candidates for standard therapy or unlikely to tolerate or derive significant clinical benefit from standard therapy, or
* has declined standard therapy

Secondary AML (MDS-related/ therapy- induced), or

Acute promyelocytic leukemia not eligible for standard therapy and/or specific therapy.

* Adequate renal and hepatic functions unless clearly disease related as indicated by the following laboratory values:

  * Serum creatinine ≤1.5 x ULN;
  * Estimated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault equation);
  * Hepatic function;

    i. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN); ii. Aspartate aminotransferase (AST)
    1. ≤2.5 × ULN
    2. ≤5 × ULN for patients with liver metastases

       iii. Alanine aminotransferase (ALT)

    <!-- -->

    1. ≤2.5 × ULN
    2. ≤5 × ULN for patients with liver metastases

       iv. Alkaline phosphatase (ALP)

    1. ≤2.5 × ULN
* European Cooperative Oncology Group (ECOG) performance status 0, 1, 2 or 3
* Female patients of childbearing potential must have a negative serum pregnancy test within 3 days prior to taking their first dose of study medication. Male patients and female patients of reproductive potential must agree to practice highly effective methods of contraception (such as hormonal implants, combined oral contraceptives, injectable contraceptives, intrauterine device with hormone spirals, total sexual abstinence, vasectomy) throughout the study and for >3 months after the last dose of study medication. Female patients are considered NOT of childbearing potential if they have a history of surgical sterility or evidence of post-menopausal status defined as any of the following:

  1. Natural menopause with last menses >1 year ago
  2. Radiation induced oophorectomy with last menses >1 year ago
  3. Chemotherapy induced menopause with last menses >1 year ago

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Patients on treatment for AML (any anti-leukemic therapy including investigational agents) or treated less than 2 weeks before inclusion.
* Concurrent history of active malignancy in the past six months prior to diagnosis except for

  * basal and squamous cell carcinoma of the skin
  * in situ carcinoma of the cervix
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease et cetera) at the investigators discretion.
* Breastfeeding women
* Cardiac dysfunction as defined by:

  * myocardial infarction within the last 3 months of study entry, or
  * congestive heart failure NYHA class IV or
  * unstable angina, or
  * unstable cardiac arrhythmias
* SARS-CoV-2 infection < 7 days or Covid-19-vaccine < 7 days from study onset
* Patients with a history of non-compliance to medical regimens or who are considered unreliable with respect to compliance.
* Patients with any serious concomitant medical condition that could, in the opinion of the investigator, compromise participation in the study.
* Patients with senile dementia, mental impairment or any other psychiatric disorder that prohibits the patient from understanding and giving informed consent.
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Known hypersensitivity to study medications or its excipients.
* Any psychological, familial, sociological, and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the treatment combinations of hydroxyurea + valproic acid, and 6-mercaptopurine + valproic acid administered at established clinical doses. | Evaluation every 4th week, i.e. after each treatment cycle.
  Safety and tolerability assessed by monitoring the incidence, frequency, and severity of AEs by using CTCAE v5.0, including evaluation of the following:
  * DLTs
  * Physical examinations
  * Clinical laboratory blood samples
Preliminary efficacy of the treatment combination of hydroxyurea and valproic acid administered at established clinical doses. | Evaluation every 4th week, i.e. after each treatment cycle.
  Clinical benefit in patients receiving hydroxyurea in combination with valproic acid.
  Clinical benefit in patients receiving 6-mercaptopurine in combination with valproic acid.
  Clinical benefit, in this protocol, is defined as stable disease, partial response (decrease of bone marrow blast percentage to between 5% to 25% and decrease of pre-treatment bone marrow blast percentage by at least 50%), or better response [European Leukemia Net (ELN) 2022 response criteria in AML], and/or stable or improved ECOG performance status.
Changes in patients performance status from baseline and during the study period. | Evaluation at baseline, i.e. before onset treatment, after 4 weeks on treatment (i.e.after first cycle), and every 4th week to a total of 24 weeks. (i.e. after each treatment cycle, up to a total of 6 cycles).
  Baseline and longitudinal ECOG performance status of the patient (Eastern Cooperative Oncology Group). The ECOG performance status scale is best at 0 (fully active, able to carry on all pre-disease performance without restriction), and worst at 5 (dead).

SECONDARY OUTCOMES:
Clinical benefit. | After 3 and 6 cycles (i.e. after 3 and 6 months from the treatment onset).
  The percentage of patients with clinical benefit (as described over) in each group (A1, A2, B1, B2).
Duration of clinical benefit. | During the treatment period of 6 months, and during follow-up, up to 6 months after end treatment.
  The duration of clinical benefit (in days), in each group (A1, A2, B1, B2).
Time to progression. | From the treatment onset, during the treatment period of 6 months, and during follow-up, up to 6 months after end treatment.
  The time to progression (days), in each group (A1, A2, B1, B2).
Changes in reported Quality of Life (QoL) compared to baseline. | At baseline, i.e. before onset treatment, after 4 weeks on treatment (i.e.after first cycle), and after each treatment cycle (every 4th week).
  Use of health-related quality of life questionnaires:
  * EQ -5D-5L
  * QLQ-C30
  * NCI- PRO-CTCAE
Survival analyses, ORR. | After 3 and 6 cycles (i.e. after 3 and 6 months from the treatment onset).
  The overall response rate (ORR) defined as the percentage of patients with a response of complete remission (CR), complete remission with incomplete hematologic recovery (CRi), morphologic leukemia-free state (MLFS), partial remission (PR), or no response, all as assessed by ELN response criteria 2022, in each group (A1, A2, B1, B2).
Survival analyses, OS. | From the treatment onset, during the treatment period of 6 months, and during follow-up, up to 6 months after end-treatment.
  The overall survival (OS), in each group (A1, A2, B1, B2).
Hospitalization rate per month per patient. | Before the treatment onset, during the treatment period of 6 months, and during follow-up, up to 6 months after end treatment.
  The number of hospital admissions per month before, during, and after study investigation.
Transfusion rate per month per patient. | Before the treatment onset, during the treatment period of 6 months, and during follow-up, up to 6 months after end treatment.
  The number of blood-/platelet transfusions per month, during and after study investigation.

OTHER OUTCOMES:
Biomarkers (exploratory). | Through study completion, an average of 5 years, or prolonged if necessary.
  Detecting changes in the expression level of intracellular or extracellular signaling markers, may predict positive pharmacological activity of the investigational combinations, and therefore treatment response. These parameters are exploratory and will be measured by mass cytometry on baseline patient samples before treatment onset, and longitudinally with the treatment, sampled every 4th week.
Relation of serum concentrations of VPA to treatment response (exploratory). | Exploratory outcome, during the study period, an average of 5 years.
  Measure of VPA concentrations in serum (normal reference values: 300 - 700 µmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Tore Gjertsen, MD, PhD, Principal Investigator — Helse-Bergen HF
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data are shared with the research group to which the PI and study staff belong to. If relevant, data can be shared with the network. All data that are to be shared will be fully anonymized and followed the relevant guidelines.
Supporting Information: Study Protocol
Time Frame: During the study period.
Access Criteria: Collaboration.

REFERENCES:
- [Background] Dohner H, Wei AH, Appelbaum FR, Craddock C, DiNardo CD, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Lowenberg B. Diagnosis and management of AML in adults: 2022 recommendations from an international expert panel on behalf of the ELN. Blood. 2022 Sep 22;140(12):1345-1377. doi: 10.1182/blood.2022016867. PMID 35797463
- [Background] Lowenberg B, Downing JR, Burnett A. Acute myeloid leukemia. N Engl J Med. 1999 Sep 30;341(14):1051-62. doi: 10.1056/NEJM199909303411407. No abstract available. PMID 10502596
- [Background] Musialek MW, Rybaczek D. Hydroxyurea-The Good, the Bad and the Ugly. Genes (Basel). 2021 Jul 19;12(7):1096. doi: 10.3390/genes12071096. PMID 34356112
- [Background] Fredly H, Gjertsen BT, Bruserud O. Histone deacetylase inhibition in the treatment of acute myeloid leukemia: the effects of valproic acid on leukemic cells, and the clinical and experimental evidence for combining valproic acid with other antileukemic agents. Clin Epigenetics. 2013 Jul 30;5(1):12. doi: 10.1186/1868-7083-5-12. PMID 23898968
- [Background] Leitch C, Osdal T, Andresen V, Molland M, Kristiansen S, Nguyen XN, Bruserud O, Gjertsen BT, McCormack E. Hydroxyurea synergizes with valproic acid in wild-type p53 acute myeloid leukaemia. Oncotarget. 2016 Feb 16;7(7):8105-18. doi: 10.18632/oncotarget.6991. PMID 26812881
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Soriano AO, Yang H, Faderl S, Estrov Z, Giles F, Ravandi F, Cortes J, Wierda WG, Ouzounian S, Quezada A, Pierce S, Estey EH, Issa JP, Kantarjian HM, Garcia-Manero G. Safety and clinical activity of the combination of 5-azacytidine, valproic acid, and all-trans retinoic acid in acute myeloid leukemia and myelodysplastic syndrome. Blood. 2007 Oct 1;110(7):2302-8. doi: 10.1182/blood-2007-03-078576. Epub 2007 Jun 27. PMID 17596541
- [Background] Chateauvieux S, Morceau F, Dicato M, Diederich M. Molecular and therapeutic potential and toxicity of valproic acid. J Biomed Biotechnol. 2010;2010:479364. doi: 10.1155/2010/479364. Epub 2010 Jul 29. PMID 20798865
- [Background] Tassara M, Dohner K, Brossart P, Held G, Gotze K, Horst HA, Ringhoffer M, Kohne CH, Kremers S, Raghavachar A, Wulf G, Kirchen H, Nachbaur D, Derigs HG, Wattad M, Koller E, Brugger W, Matzdorff A, Greil R, Heil G, Paschka P, Gaidzik VI, Gottlicher M, Dohner H, Schlenk RF. Valproic acid in combination with all-trans retinoic acid and intensive therapy for acute myeloid leukemia in older patients. Blood. 2014 Jun 26;123(26):4027-36. doi: 10.1182/blood-2013-12-546283. Epub 2014 May 5. PMID 24797300
- [Background] Elion GB. Historical background of 6-mercaptopurine. Toxicol Ind Health. 1986 Sep;2(2):1-9. doi: 10.1177/074823378600200201. No abstract available. PMID 3538499
- [Background] BURCHENAL JH, MURPHY ML, ELLISON RR, SYKES MP, TAN TC, LEONE LA, KARNOFSKY DA, CRAVER LF, DARGEON HW, RHOADS CP. Clinical evaluation of a new antimetabolite, 6-mercaptopurine, in the treatment of leukemia and allied diseases. Blood. 1953 Nov;8(11):965-99. No abstract available. PMID 13105700
- [Background] Burnett A, Wetzler M, Lowenberg B. Therapeutic advances in acute myeloid leukemia. J Clin Oncol. 2011 Feb 10;29(5):487-94. doi: 10.1200/JCO.2010.30.1820. Epub 2011 Jan 10. PMID 21220605
- [Background] Estey E. Acute myeloid leukemia and myelodysplastic syndromes in older patients. J Clin Oncol. 2007 May 10;25(14):1908-15. doi: 10.1200/JCO.2006.10.2731. PMID 17488990
- [Background] Hiddemann W, Kern W, Schoch C, Fonatsch C, Heinecke A, Wormann B, Buchner T. Management of acute myeloid leukemia in elderly patients. J Clin Oncol. 1999 Nov;17(11):3569-76. doi: 10.1200/JCO.1999.17.11.3569. PMID 10550156
- [Background] Kantarjian HM, Thomas XG, Dmoszynska A, Wierzbowska A, Mazur G, Mayer J, Gau JP, Chou WC, Buckstein R, Cermak J, Kuo CY, Oriol A, Ravandi F, Faderl S, Delaunay J, Lysak D, Minden M, Arthur C. Multicenter, randomized, open-label, phase III trial of decitabine versus patient choice, with physician advice, of either supportive care or low-dose cytarabine for the treatment of older patients with newly diagnosed acute myeloid leukemia. J Clin Oncol. 2012 Jul 20;30(21):2670-7. doi: 10.1200/JCO.2011.38.9429. Epub 2012 Jun 11. PMID 22689805
- [Background] Wei AH, Panayiotidis P, Montesinos P, Laribi K, Ivanov V, Kim I, Novak J, Stevens DA, Fiedler W, Pagoni M, Bergeron J, Ting SB, Hou JZ, Anagnostopoulos A, McDonald A, Murthy V, Yamauchi T, Wang J, Chyla B, Sun Y, Jiang Q, Mendes W, Hayslip J, DiNardo CD. 6-month follow-up of VIALE-C demonstrates improved and durable efficacy in patients with untreated AML ineligible for intensive chemotherapy (141/150). Blood Cancer J. 2021 Oct 1;11(10):163. doi: 10.1038/s41408-021-00555-8. PMID 34599139
- [Background] Pollyea DA, DiNardo CD, Arellano ML, Pigneux A, Fiedler W, Konopleva M, Rizzieri DA, Smith BD, Shinagawa A, Lemoli RM, Dail M, Duan Y, Chyla B, Potluri J, Miller CL, Kantarjian HM. Impact of Venetoclax and Azacitidine in Treatment-Naive Patients with Acute Myeloid Leukemia and IDH1/2 Mutations. Clin Cancer Res. 2022 Jul 1;28(13):2753-2761. doi: 10.1158/1078-0432.CCR-21-3467. PMID 35046058
- [Background] Steensma DP, Tefferi A. The myelodysplastic syndrome(s): a perspective and review highlighting current controversies. Leuk Res. 2003 Feb;27(2):95-120. doi: 10.1016/s0145-2126(02)00098-x. PMID 12526916
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Catenacci DV, Schiller GJ. Myelodysplasic syndromes: a comprehensive review. Blood Rev. 2005 Nov;19(6):301-19. doi: 10.1016/j.blre.2005.01.004. PMID 15885860
- [Background] Greenberg PL, Stone RM, Al-Kali A, Barta SK, Bejar R, Bennett JM, Carraway H, De Castro CM, Deeg HJ, DeZern AE, Fathi AT, Frankfurt O, Gaensler K, Garcia-Manero G, Griffiths EA, Head D, Horsfall R, Johnson RA, Juckett M, Klimek VM, Komrokji R, Kujawski LA, Maness LJ, O'Donnell MR, Pollyea DA, Shami PJ, Stein BL, Walker AR, Westervelt P, Zeidan A, Shead DA, Smith C. Myelodysplastic Syndromes, Version 2.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Jan;15(1):60-87. doi: 10.6004/jnccn.2017.0007. PMID 28040720
- [Background] Lubbert M. DNA methylation inhibitors in the treatment of leukemias, myelodysplastic syndromes and hemoglobinopathies: clinical results and possible mechanisms of action. Curr Top Microbiol Immunol. 2000;249:135-64. doi: 10.1007/978-3-642-59696-4_9. No abstract available. PMID 10802943
- [Background] Pfeilstocker M, Tuechler H, Sanz G, Schanz J, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Levis A, Luebbert M, Maciejewski J, Machherndl-Spandl S, Magalhaes SM, Miyazaki Y, Sekeres MA, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D, Greenberg PL. Time-dependent changes in mortality and transformation risk in MDS. Blood. 2016 Aug 18;128(7):902-10. doi: 10.1182/blood-2016-02-700054. Epub 2016 Jun 22. PMID 27335276
- [Background] Rowley JD, Golomb HM, Dougherty C. 15/17 translocation, a consistent chromosomal change in acute promyelocytic leukaemia. Lancet. 1977 Mar 5;1(8010):549-50. doi: 10.1016/s0140-6736(77)91415-5. No abstract available. PMID 65649
- [Background] Grignani F, Ferrucci PF, Testa U, Talamo G, Fagioli M, Alcalay M, Mencarelli A, Grignani F, Peschle C, Nicoletti I, et al. The acute promyelocytic leukemia-specific PML-RAR alpha fusion protein inhibits differentiation and promotes survival of myeloid precursor cells. Cell. 1993 Aug 13;74(3):423-31. doi: 10.1016/0092-8674(93)80044-f. PMID 8394219
- [Background] Lo-Coco F, Cicconi L. History of acute promyelocytic leukemia: a tale of endless revolution. Mediterr J Hematol Infect Dis. 2011;3(1):e2011067. doi: 10.4084/MJHID.2011.067. Epub 2011 Dec 21. No abstract available. PMID 22220264
- [Background] Breitman TR, Selonick SE, Collins SJ. Induction of differentiation of the human promyelocytic leukemia cell line (HL-60) by retinoic acid. Proc Natl Acad Sci U S A. 1980 May;77(5):2936-40. doi: 10.1073/pnas.77.5.2936. PMID 6930676
- [Background] Park JH, Qiao B, Panageas KS, Schymura MJ, Jurcic JG, Rosenblat TL, Altman JK, Douer D, Rowe JM, Tallman MS. Early death rate in acute promyelocytic leukemia remains high despite all-trans retinoic acid. Blood. 2011 Aug 4;118(5):1248-54. doi: 10.1182/blood-2011-04-346437. Epub 2011 Jun 8. PMID 21653939
- [Background] Mantha S, Tallman MS, Devlin SM, Soff GA. Predictive factors of fatal bleeding in acute promyelocytic leukemia. Thromb Res. 2018 Apr;164 Suppl 1:S98-S102. doi: 10.1016/j.thromres.2018.01.038. PMID 29703492
- [Background] Abaza Y, Kantarjian H, Garcia-Manero G, Estey E, Borthakur G, Jabbour E, Faderl S, O'Brien S, Wierda W, Pierce S, Brandt M, McCue D, Luthra R, Patel K, Kornblau S, Kadia T, Daver N, DiNardo C, Jain N, Verstovsek S, Ferrajoli A, Andreeff M, Konopleva M, Estrov Z, Foudray M, McCue D, Cortes J, Ravandi F. Long-term outcome of acute promyelocytic leukemia treated with all-trans-retinoic acid, arsenic trioxide, and gemtuzumab. Blood. 2017 Mar 9;129(10):1275-1283. doi: 10.1182/blood-2016-09-736686. Epub 2016 Dec 21. PMID 28003274
- [Background] Iland HJ, Collins M, Bradstock K, Supple SG, Catalano A, Hertzberg M, Browett P, Grigg A, Firkin F, Campbell LJ, Hugman A, Reynolds J, Di Iulio J, Tiley C, Taylor K, Filshie R, Seldon M, Taper J, Szer J, Moore J, Bashford J, Seymour JF; Australasian Leukaemia and Lymphoma Group. Use of arsenic trioxide in remission induction and consolidation therapy for acute promyelocytic leukaemia in the Australasian Leukaemia and Lymphoma Group (ALLG) APML4 study: a non-randomised phase 2 trial. Lancet Haematol. 2015 Sep;2(9):e357-66. doi: 10.1016/S2352-3026(15)00115-5. Epub 2015 Aug 20. PMID 26685769
- [Background] Tallman MS, Andersen JW, Schiffer CA, Appelbaum FR, Feusner JH, Woods WG, Ogden A, Weinstein H, Shepherd L, Willman C, Bloomfield CD, Rowe JM, Wiernik PH. All-trans retinoic acid in acute promyelocytic leukemia: long-term outcome and prognostic factor analysis from the North American Intergroup protocol. Blood. 2002 Dec 15;100(13):4298-302. doi: 10.1182/blood-2002-02-0632. Epub 2002 Aug 15. PMID 12393590
- [Background] Dresler WFC, Stein R. Über den hydroxylharnstoff. Justus Liebigs Ann Chem. 1869;150:242- 52. https://doi.org/10.1002/jlac.18691500212.
- [Background] Lancet JE, Moseley A, Komrokji RS, Coutre SE, DeAngelo DJ, Tallman MS, Litzow M, Othus M, Appelbaum FR. ATRA, Arsenic Trioxide (ATO), and Gemtuzumab Ozogamicin (GO) Is Safe and Highly Effective in Patients with Previously Untreated High-Risk Acute Promyelocytic Leukemia (APL): Final Results of the SWOG/Alliance/ ECOG S0535 Trial. Blood. 2016; 128:896. https://doi. org/10.1182/blood.V128.22.896.896
- [Background] Rosenthal F, Wislicki L, Kollek L: Über die Beziehungen von schwersten Blutgiften zu Abbauproducten des Eiweisses: ein Beitrag zum Einstehungsmechanismus der perniziösen änamie. Klin Wochenschr 7:972-977, 1928
- [Background] STEARNS B, LOSEE KA, BERNSTEIN J. HYDROXYUREA. A NEW TYPE OF POTENTIAL ANTITUMOR AGENT. J Med Chem. 1963 Mar;6:201. doi: 10.1021/jm00338a026. No abstract available. PMID 14188794
- [Background] Gwilt PR, Tracewell WG. Pharmacokinetics and pharmacodynamics of hydroxyurea. Clin Pharmacokinet. 1998 May;34(5):347-58. doi: 10.2165/00003088-199834050-00002. PMID 9592619
- [Background] Leavell UW Jr, Yarbro JW. Hydroxyurea. A new treatment for psoriasis. Arch Dermatol. 1970 Aug;102(2):144-50. doi: 10.1001/archderm.102.2.144. No abstract available. PMID 4914264
- [Background] Cannas G, Poutrel S, Thomas X. Hydroxycarbamine: from an Old Drug Used in Malignant Hemopathies to a Current Standard in Sickle Cell Disease. Mediterr J Hematol Infect Dis. 2017 Feb 15;9(1):e2017015. doi: 10.4084/MJHID.2017.015. eCollection 2017. PMID 28293403
- [Background] BS B. On the propyl derivatives and decomposition products of ethylacetoacetate. Am Chem J 1882;3:385-395.
- [Background] MEUNIER H, CARRAZ G, NEUNIER Y, EYMARD P, AIMARD M. [Pharmacodynamic properties of N-dipropylacetic acid]. Therapie. 1963 Mar-Apr;18:435-8. No abstract available. French. PMID 13935231
- [Background] Gottlicher M, Minucci S, Zhu P, Kramer OH, Schimpf A, Giavara S, Sleeman JP, Lo Coco F, Nervi C, Pelicci PG, Heinzel T. Valproic acid defines a novel class of HDAC inhibitors inducing differentiation of transformed cells. EMBO J. 2001 Dec 17;20(24):6969-78. doi: 10.1093/emboj/20.24.6969. PMID 11742974
- [Background] Chen Y, Tsai YH, Tseng SH. Combined valproic acid and celecoxib treatment induced synergistic cytotoxicity and apoptosis in neuroblastoma cells. Anticancer Res. 2011 Jun;31(6):2231-9. PMID 21737646
- [Background] Das CM, Aguilera D, Vasquez H, Prasad P, Zhang M, Wolff JE, Gopalakrishnan V. Valproic acid induces p21 and topoisomerase-II (alpha/beta) expression and synergistically enhances etoposide cytotoxicity in human glioblastoma cell lines. J Neurooncol. 2007 Nov;85(2):159-70. doi: 10.1007/s11060-007-9402-7. Epub 2007 May 30. PMID 17534580
- [Background] McCormack E, Haaland I, Venas G, Forthun RB, Huseby S, Gausdal G, Knappskog S, Micklem DR, Lorens JB, Bruserud O, Gjertsen BT. Synergistic induction of p53 mediated apoptosis by valproic acid and nutlin-3 in acute myeloid leukemia. Leukemia. 2012 May;26(5):910-7. doi: 10.1038/leu.2011.315. Epub 2011 Nov 8. PMID 22064349
- [Background] Steinberg MH, McCarthy WF, Castro O, Ballas SK, Armstrong FD, Smith W, Ataga K, Swerdlow P, Kutlar A, DeCastro L, Waclawiw MA; Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell Anemia and MSH Patients' Follow-Up. The risks and benefits of long-term use of hydroxyurea in sickle cell anemia: A 17.5 year follow-up. Am J Hematol. 2010 Jun;85(6):403-8. doi: 10.1002/ajh.21699. PMID 20513116
- [Background] Hankins JS, Aygun B, Nottage K, Thornburg C, Smeltzer MP, Ware RE, Wang WC. From infancy to adolescence: fifteen years of continuous treatment with hydroxyurea in sickle cell anemia. Medicine (Baltimore). 2014 Dec;93(28):e215. doi: 10.1097/MD.0000000000000215. PMID 25526439
- [Background] Fredly H, Stapnes Bjornsen C, Gjertsen BT, Bruserud O. Combination of the histone deacetylase inhibitor valproic acid with oral hydroxyurea or 6-mercaptopurin can be safe and effective in patients with advanced acute myeloid leukaemia--a report of five cases. Hematology. 2010 Oct;15(5):338-43. doi: 10.1179/102453310X12647083620967. PMID 20863429
- [Background] Andresen V, Gjertsen BT. Drug Repurposing for the Treatment of Acute Myeloid Leukemia. Front Med (Lausanne). 2017 Nov 29;4:211. doi: 10.3389/fmed.2017.00211. eCollection 2017. PMID 29238707
- [Background] Jadersten M, Lilienthal I, Tsesmetzis N, Lourda M, Bengtzen S, Bohlin A, Arnroth C, Erkers T, Seashore-Ludlow B, Giraud G, Barkhordar GS, Tao S, Fogelstrand L, Saft L, Ostling P, Schinazi RF, Kim B, Schaller T, Juliusson G, Deneberg S, Lehmann S, Rassidakis GZ, Hoglund M, Henter JI, Herold N. Targeting SAMHD1 with hydroxyurea in first-line cytarabine-based therapy of newly diagnosed acute myeloid leukaemia: Results from the HEAT-AML trial. J Intern Med. 2022 Dec;292(6):925-940. doi: 10.1111/joim.13553. Epub 2022 Aug 18. PMID 35934913
- [Background] Mamez AC, Raffoux E, Chevret S, Lemiale V, Boissel N, Canet E, Schlemmer B, Dombret H, Azoulay E, Lengline E. Pre-treatment with oral hydroxyurea prior to intensive chemotherapy improves early survival of patients with high hyperleukocytosis in acute myeloid leukemia. Leuk Lymphoma. 2016 Oct;57(10):2281-8. doi: 10.3109/10428194.2016.1142083. Epub 2016 Feb 5. PMID 26849624
- [Background] Grund FM, Armitage JO, Burns P. Hydroxyurea in the prevention of the effects of leukostasis in acute leukemia. Arch Intern Med. 1977 Sep;137(9):1246-7. PMID 268956
- [Background] Berg J, Vincent PC, Gunz FW. Extreme leucocytosis and prognosis of newly diagnosed patients with acute non-lymphocytic leukaemia. Med J Aust. 1979 Jun 2;1(11):480-2. doi: 10.5694/j.1326-5377.1979.tb119318.x. PMID 288967
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Fredly H, Ersvaer E, Kittang AO, Tsykunova G, Gjertsen BT, Bruserud O. The combination of valproic acid, all-trans retinoic acid and low-dose cytarabine as disease-stabilizing treatment in acute myeloid leukemia. Clin Epigenetics. 2013 Aug 1;5(1):13. doi: 10.1186/1868-7083-5-13. PMID 23915396
- [Background] Kuendgen A, Strupp C, Aivado M, Bernhardt A, Hildebrandt B, Haas R, Germing U, Gattermann N. Treatment of myelodysplastic syndromes with valproic acid alone or in combination with all-trans retinoic acid. Blood. 2004 Sep 1;104(5):1266-9. doi: 10.1182/blood-2003-12-4333. Epub 2004 May 20. PMID 15155466
- [Background] Raffoux E, Chaibi P, Dombret H, Degos L. Valproic acid and all-trans retinoic acid for the treatment of elderly patients with acute myeloid leukemia. Haematologica. 2005 Jul;90(7):986-8. PMID 15996941
- [Background] STOCK CC, CLARKE DA, PHILIPS FS, BARCLAY RK, MYRON SA. Sarcoma 180 screening data. Cancer Res. 1960 Jun;20(5)Pt 2:193-381. No abstract available. PMID 13834725
- See also: The Nobel Prize in Physiology or Medicine 1988 was awarded jointly to Sir James W. Black, Gertrude B. Elion and George H. Hitchings for their discoveries of important principles for drug treatment. — https://www.nobelprize.org/prizes/medicine/1988/summary/
- See also: Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia — http://pubmed.ncbi.nlm.nih.gov/32786187/
- See also: Sarcoma 180 screening data — https://www.abcam.com/hydroxyurea-colorimetric-assay-kit-ab282919.html